CLINICAL TRIAL: NCT01612143
Title: A Randomized, Open-label, Single Dose, Cross-over Study to Investigate the Relative Bioavailability of Setrobuvir (STV) Tablet Formulation Versus the Reference Setrobuvir Capsule Formulation Following Oral Administration With or Without a High Fat Meal in Healthy Subjects
Brief Title: A Relative Bioavailability Study of Setrobuvir Tablet Formulation Versus Reference Setrobuvir Capsule Formulation in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: NP28327; 2012-001001-24 (EudraCT Number)
Record Dates: First submitted 2012-06-01; First posted 2012-06-05 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — setrobuvir

ARMS (4):
- A: STV capsule (after high fat meal) (Active Comparator)
  Interventions: Drug: setrobuvir
- B: STV capsule (fasted state) (Active Comparator)
  Interventions: Drug: setrobuvir
- C: STV tablet (after high fat meal) (Experimental)
  Interventions: Drug: setrobuvir
- D: STV tablet (fasted state) (Experimental)
  Interventions: Drug: setrobuvir

INTERVENTIONS:
Drug: setrobuvir — 200 mg capsule formulation, single oral dose
  Arms: A: STV capsule (after high fat meal); B: STV capsule (fasted state)
Drug: setrobuvir — 200 mg tablet formulation, single oral dose
  Arms: C: STV tablet (after high fat meal); D: STV tablet (fasted state)

SUMMARY:
This open-label, randomized, single dose, 4-sequence, 4-period crossover study will assess the relative bioavailability of setrobuvir as tablet formulation versus the reference capsule formulation in healthy volunteers. Subjects will be randomized to one of four treatment sequences receiving 4 single oral doses of 200 mg setrobuvir, either as tablet or capsule formulation with or without a high fat meal, with a washout period of at least 14 days between treatments.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female adults, 18 to 55 years of age inclusive
* Body mass index (BMI) 18.0 - 30.0 kg/m2
* Healthy status defined as absence of clinically significant acute or chronic condition as determined by complete medical history and physical examination
* Females of childbearing potential and males and their female partner(s) of childbearing potential must agree to use 2 forms of contraception as defined by protocol during treatment and for at least 3 months after the last dose of study drug
* Non-smokers or use of < 10 cigarettes (or equivalent nicotine-containing product) per day
* Negative results on following screening laboratory test: urine drug screen, urine alcohol screen
* Willing and able to consume the study-specified meal on day of dosing

Exclusion Criteria:

* Pregnant or lactating women, or males with female partners who are pregnant or lactating
* History of current alcohol abuse and/or other drug addiction </= 2 years prior to enrollment in the study
* Participation in other clinical studies within 60 days prior to study randomization
* Positive for hepatitis B, hepatitis C or HIV infection

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2012-06; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Relative bioavailability: Cmax/area under the concentration-time curve (AUC) | Pre-dose and up to 168 hours post-dose

SECONDARY OUTCOMES:
Safety: Incidence of adverse events | approximately 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Zuidlaren, Netherlands